CLINICAL TRIAL: NCT01367145
Title: OMEGA-3-POLYUNSATURATED FATTY-ACIDS (n3-PUFA) IN PATIENTS WITH PERIPHERAL ARTERIAL DISEASE: EFFECTS ON ENDOTHELIAL FUNCTION - A RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND TRIAL
Brief Title: OMEGA-3-Polyunsaturated Fatty-Acids (N3-Pufa) In Patients With Peripheral Arterial Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sabine Steiner, Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OMACOR II - 2011
Record Dates: First submitted 2011-05-09; First posted 2011-06-06 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Peripheral Arterial Disease
Keywords: OMEGA-3 polyunsaturated fatty-acids; Peripheral Arterial Disease; Endothelial Function; Inflammation; Platelet Function
MeSH Terms: conditions — Peripheral Arterial Disease; Inflammation | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omacor (Active Comparator)
  Interventions: Drug: OMACOR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMACOR — 4 capsules OMACOR 1g per day
  Arms: Omacor
Drug: Placebo — 4 capsules placebo per day
  Arms: Placebo

SUMMARY:
The principal aim of the study is to determine the effects n3-PUFA on top of standard therapy on surrogate markers of disease severity and/or prognosis in patients with PAD.

Treatment duration will be 3 months, final follow-up is planned at 6 months after inclusion.

Primary outcome parameter is endothelial function assessed by flow-mediated vasodilation using brachial artery ultrasound.

Secondary outcome measures comprise maximum and pain-free treadmill walking distance, pulse wave velocity, whole blood viscosity, platelet activation and plasma markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Severity of disease: Rutherford category II or III - moderate to severe Stable intermittent claudication
* Ankle Brachial Index<0.9
* Age ≥18 years
* Adequate PAD therapy according to current AHA guidelines

Exclusion Criteria:

* Current treatment with Omacor or other fish oil products
* Planned vascular intervention
* Known hypersensitivity to the study drug
* Rest pain or ischemic ulcer
* Exercise tolerance limited by factors other than PAD
* Inability to perform treadmill test
* Dual antiplatelet therapy (aspirin and clopidogrel)
* Previous myocardial infarction
* Known liver diseases, except fatty liver
* Known bleeding diathesis
* Women of childbearing potential who do not practice a safe contraception method
* Current participation in another intervention study.
* Previous participation in another study with an intervention within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change from baseline endothelial function to 3 months | baseline, 3 months
  measured by flow mediated vasodilation

SECONDARY OUTCOMES:
change from baseline endothelial function to six months | baseline, 6 months (3 months after treatment cessation)
change of walking distance (maximum/pain-free)from baseline to three months and six months | baseline, 3, 6 months
change of inflammatory markers from baseline to one, three and six months | baseline, 1, 3, 6 months
change of pulse wave velocity from baseline to one, three and six months | baseline, 1, 3, 6 months
bleeding events | 1, 3, 6 months
liver enzymes changes | baseline, 1,3,6 months
change of platelet activation from baseline to one, three and six months | baseline, 1, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Steiner, Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Internal Medicine II, Division of Angiology, Vienna, Austria